CLINICAL TRIAL: NCT00734851
Title: Multimodality Therapy for Recurrent High Risk Prostate Cancer: A Phase II Study
Brief Title: Multimodality Phase II Study in Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Dose Limiting Toxicities
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010747
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; sunitinib; docetaxel; PSA; radiation; PSA recurrence; No metastatic disease
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multimodality (Experimental): 4 cycles of 70 mg/m2 Docetaxel + 37.5 mg daily Sunitinib for 14 days followed by a 7 day break for 3 cycles + external beam radiotherapy to 66 Gray over 6-7 weeks
  Interventions: Drug: Docetaxel; Drug: Sunitinib; Radiation: EBXRT

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 70 mg/m2 day 1 every 3 weeks for 4 cycles with prednisone 5 mg orally twice daily
  Other Names: Taxotere
Drug: Sunitinib — Sunitinib 37.5 mg orally once daily for 14 days followed by 7 days off, for 4 cycles, concurrent with docetaxel and prednisone
  Other Names: Sutent
Radiation: EBXRT — External beam radiotherapy to the prostate bed, started on day 100, after completion of chemotherapy. 66 Gy over 6-7 weeks.
  Other Names: IMRT

SUMMARY:
This is a single arm phase II study of docetaxel, prednisone, and sunitinib systemic therapy followed by salvage external beam radiation therapy for men who have experienced PSA recurrence following initial radical prostatectomy for prostate cancer. The primary aim is the rate of progression-free survival at 2 years as measured by lack of PSA progression and no evidence of disease. We hypothesize that this aggressive initial systemic therapy will improve the long term remission rates for men who are undergoing salvage radiation therapy for PSA recurrence in the absence of metastatic disease.

DETAILED DESCRIPTION:
In many common malignancies such as breast cancer, trimodality therapy represents the standard-of-care approach, including initial surgical resection followed by systemic chemotherapy followed by radiotherapy for optimal local control, and targeted hormonal or biologic therapy for a period of time to reduce the ongoing risk of systemic disease recurrence. These approaches have reduced recurrence rates and improved overall survival in the adjuvant setting in breast cancer; however, the treatment of men with PSA recurrence following radical prostatectomy has generally been unsatisfying, given the high rates of persistent or recurrent disease despite salvage radiotherapy.

The primary purpose of the study is to determine the rate of biochemical (PSA) progression free survival (bPFS) in men with PSA recurrent non-metastatic prostate cancer following radical prostatectomy, who receive multimodality therapy consisting of local salvage external beam radiotherapy and systemic docetaxel-based chemotherapy plus the targeted anti-VEGF biologic therapy sunitinib. Biochemical PFS will be defined as the proportion of subjects at 24 months, post-registration, with one of the following: 1) a serum PSA value of 0.2 ng/ml or more above the post-radiotherapy PSA nadir and confirmed 4 weeks later by a second PSA measurement that was higher than the first by any amount, 2) a continued rise in the PSA level following study treatment if no nadir is experienced, defined as 2 rising values greater than the baseline PSA and separated by at least 4 weeks, 3) evidence of clinical progression or initiation of systemic therapy for progressive disease, or 4) death. Secondary objectives include finding the rate of biochemical (PSA) disease free survival over time, Two-, three-, five-, and six- year risk of local recurrence (proportion), two-, three-, five-, and six-year risk of metastases and metastasis-free survival, two-, three-, five-, and six-year risk of metastases and metastasis-free survival, Safety, feasibility, and tolerability as assessed by NCI Common Toxicity Scales (v3.0), quality of life questionnaire (EPIC-short form surveys), achievement of accrual goals. Finally, a comparison of RNA expression profiles from original prostate radical prostatectomy specimen among those with PSA relapse at 2 and 5 years as compared to those without PSA relapse at the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Prostate adenocarcinoma with evidence of recurrent disease as measured only by rising PSA, without evidence of metastatic disease by bone scan or CT scan within 4 weeks of entry
2. PSA ≤ 3.0 ng/ml and ≥ 0.1 ng/ml within 2 weeks of registration
3. Radical prostatectomy within 4 years of registration.
4. Rising PSA as defined by 1 or more PSA values greater than the nadir value after radical prostatectomy, separated by at least 4 weeks.
5. Gleason sum at radical prostatectomy of 7-10 (4+3 or 3+4 allowed)
6. Informed consent
7. Age > 18 years.
8. Adequate laboratory parameters:

   * leukocytes ≥ 3,000/uL
   * absolute neutrophil count ≥ 1,500/uL
   * platelets ≥ 75,000/uL
   * hemoglobin > 9.0 g/dl
   * total bilirubin within normal institutional limit
   * AST(SGOT)/ALT(SGPT) < 2.5x institutional upper limit
   * creatinine < 2.0x institutional upper limit
9. Karnofsky Performance Status ≥ 80 (Attachment 2).
10. Written, signed, dated, and witnessed IRB approved informed consent form (ICF) before any screening procedures are performed.
11. Peripheral neuropathy ≤ grade 1

Exclusion Criteria:

1. Evidence of metastatic disease by CT scan, physical exam, or bone scan within 4 weeks of registration
2. History of bleeding disorders or medical comorbidities that in the opinion of the investigator would preclude the use of systemic chemotherapy
3. Prior systemic or biologic therapy, including pre-operative therapies or adjuvant chemotherapy, biologic therapy, or hormonal therapy
4. Life expectancy of less than 5 years from medical co-morbidities by physician judgment
5. Non-adenocarcinoma prostate cancer pathology at radical prostatectomy
6. Prior radiotherapy to the abdomen or pelvis
7. Less than or equal to 6 weeks from prior major surgery, including radical prostatectomy, open biopsy, or traumatic injury.
8. Recent cardiovascular event (within 12 months) including unstable angina, myocardial infarction, severe or at rest claudication, or stroke/CVA.
9. Subjects receiving known strong CYP3A4 isoenzyme inhibitors and/or inducers. Subjects on acceptable CYP3A4 isoenzyme inhibitors and/or inducers are eligible, provided they have been taking a stable regimen for at least 4 weeks prior to screening.
10. Presence of a non-healing wound or ulcer.
11. Grade >= 3 hemorrhage within the past month.
12. Hypertension with systolic blood pressure of >140 mm Hg and/or diastolic pressure >90 mm Hg at the time of screening. Anti-hypertensive medications are permitted.
13. Subjects with American Heart Association (AHA) Class 2-4 heart disease or any history of congestive heart failure with an ejection fraction <50%.
14. Subjects with inability to tolerate or absorb oral medications.
15. QTc interval >480 msec on baseline EKG. Subjects may not be taking a medication known to significantly prolong the QTc interval.
16. Subjects who have not recovered from prior biopsy, surgery, traumatic injury, and/or radiation therapy.
17. Anticoagulation with warfarin (therapeutic doses of warfarin for catheter patency are permitted). Low molecular weight heparin is permitted.
18. Active infection(s), active antimicrobial therapy or serious intercurrent illness.
19. Any other major medical or psychiatric illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study, including inability to absorb oral medications.
20. Any history of hemoptysis within the past 12 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-12; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Armstrong, MD, ScM, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 36 participants consented. 2 participants withdrew consent prior to going on treatment. 34 participants started treatment. 2 participants withdrew while on treatment. 18 withdrawn by PI.
Period: Overall Study
Arm/Group | Multimodality
Started | 34
Completed | 13
Not Completed | 21
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 18

BASELINE CHARACTERISTICS:
Arm/Group | Multimodality
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.76 (7.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Progression Free Survival (PFS) at 24 Months
Description: Percentage of participants surviving 24 months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression. Progression will be defined as having experienced any of the following: a serum prostate specific antigen (PSA) value of 0.2 ng/mL or more above the post-radiotherapy PSA nadir and confirmed 4 weeks later by a second PSA measurement that was higher than the first by any amount, a continued rise in the PSA level following study treatment if no nadir is experienced, defined as 2 rising values greater than the baseline PSA and separated by at least 4 weeks, or evidence of clinical progression or initiation of systemic therapy for progressive disease.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Multimodality
Number analyzed (Participants) | 34
percentage of patients | 51 [33 to 67]

2. Secondary Outcome: Proportion of Biochemical Progression (bPFS Proportion) at 2 and 3 Years.
Description: Percentage of participants surviving 24 and 36 months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression. Progression will be defined as having experienced any of the following: a serum prostate specific antigen (PSA) value of 0.2 ng/mL or more above the post-radiotherapy PSA nadir and confirmed 4 weeks later by a second PSA measurement that was higher than the first by any amount or a continued rise in the PSA level following study treatment if no nadir is experienced, defined as 2 rising values greater than the baseline PSA and separated by at least 4 weeks. Please note: bPFS is identical to PFS but includes only PSA-based endpoints or death.
Time Frame: 24 months and 36 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Multimodality
Number analyzed (Participants) | 34
percentage of patients
  24 Months | 51 [33 to 67]
  36 Months | 48 [29 to 64]

3. Secondary Outcome: Rate of Local Recurrence at 2 and 3 Years
Description: Local recurrence is defined as men with locally recurrent disease confirmed pathologically within the radiation field, and is estimated at 2 and 3 years.
Time Frame: 24 months and 36 months
Measure: Number; unit: percentage of participants
Arm/Group | Multimodality
Number analyzed (Participants) | 34
percentage of participants
  24 Months | 0
  36 Months | 0

4. Secondary Outcome: Metastasis-free Survival (MFS) Rates at 2 and 3 Years.
Description: MFS is defined as the length of time between the date of start of treatment and the date of evidence of systemic disease on bone scan or cross sectional imaging or death, whichever occurs first.
Time Frame: 2 and 3 years
Population: This rate is not estimable as 0 patients had locally recurrent disease before being taken off study for biochemical progression.
Arm/Group | Multimodality
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Quality of Life (QoL) After 1 Year
Description: A validated scale of prostate-cancer specific quality of life will be measured using the Expanded Prostate Cancer Index Composite (EPIC) short form survey. This survey is standardized into subscale, 4 of which were examined on this study. These subscales are the urinary irritative domain, urinary incontinence domain, bowel domain, and sexual function domain, each standardized on a scale of 0-100, where higher score indicate a higher level of QoL. The survey was performed at baseline, at 3 months after completing radiotherapy, at 12 months, and at 2 and 3 years of follow-up for a total of 5 possible surveys per patient. Due to a low number of completed surveys at the fourth and fifth time point, the difference between the 12 month time point and baseline is summarized. Negative values indicate a decrease in QoL, while positive numbers represent an increase.
Time Frame: baseline and 1 year
Population: Only participant who adequately completed the sub-section of each questionnaire are included in the analysis population. Some participants did not answer a sufficient number of questions to adequately score a domain and therefore were not included.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Multimodality
Number analyzed (Participants) | 21
units on a scale
  Urinary Irritative (N=20) | 0 [-75 to 12.5]
  Urinary Incontinence (N=21) | 0 [-91.75 to 29]
  Bowel (N=19) | 0 [-50 to 29.17]
  Sexual (N=21) | 0 [-12.5 to 63.83]

6. Secondary Outcome: Change in Quality of Life (QoL) After 3 Month
Description: A validated scale of prostate-cancer specific quality of life will be measured using the Expanded Prostate Cancer Index Composite (EPIC) short form survey. This survey is standardized into subscale, 4 of which were examined on this study. These subscales are the urinary irritative domain, urinary incontinence domain, bowel domain, and sexual function domain, each standardized on a scale of 0-100, where higher score indicate a higher level of QoL. The survey was performed at baseline and 3 months after completing radiotherapy. Negative values indicate a decrease in QoL, while positive numbers represent an increase.
Time Frame: baseline and 3 months
Population: as for outcome 5
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Multimodality
Number analyzed (Participants) | 32
units on a scale
  Urinary Irritative (N=29) | 0 [-25 to 43.75]
  Urinary Incontinence (N=31) | -6 [-25 to 25.25]
  Bowel (N=32) | 0 [-29.17 to 24.17]
  Sexual (N=30) | 0 [-37.5 to 26.33]

7. Secondary Outcome: Comparison of RNA Expression Profile From Original Prostate Radical Prostatectomy Specimen Among Those With PSA Relapse at 2 and 3 Years as Compared to Those Without PSA Relapse at the Primary Endpoint.
Description: Prospective collection of prostate tissue at the time of radical prostatectomy is routinely performed at Duke. These samples will be analyzed by laser capture microdissection (LCM) for genomic profiling by RNA expression analysis for all subjects with tissue available. The expression profiles of subjects who experience PSA recurrence after protocol therapy by the 24 month endpoint will be compared with the expression profiles of subjects without recurrence at this time point as an exploratory measure to predict aggressive prostate cancer and those subjects who are unlikely to benefit from this approach. Baseline prostate tumor biomarkers in the form of RNA expression profiles will be correlated with 2 year PFS in an exploratory analysis. The median bPFS of those with detectable biomarker expression is reported.
Time Frame: 2 and 3 years
Population: Due to the unavailability of tissue, this outcome was not performed.
Arm/Group | Multimodality
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 36 Months
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.3.0, and have been converted to v.4.0 for entry into ClinicalTrials.gov
Arm/Group | Multimodality
Serious Adverse Events (participants affected / at risk) | 7/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multimodality (N=34)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Lung infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multimodality (N=34)
Anemia (Blood and lymphatic system disorders) | 5
Hemolysis (Blood and lymphatic system disorders) | 1
Ear and labyrinth disorders - Other, specify: Ear Wax (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 2
Dry eye (Eye disorders) | 1
Extraocular muscle paresis (Eye disorders) | 1
Watering eyes (Eye disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Anal mucositis (Gastrointestinal disorders) | 2
Anal pain (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 24
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 14
Dysphagia (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify: Blood in stool (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: GERD (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Indigestion (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Mouth sensitivity (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: intermittent bloody stoo (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: stomach ache (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 13
Oral pain (Gastrointestinal disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 31
Fever (General disorders) | 7
General disorders and administration site conditions - Other, specify (General disorders) | 1
Pain (General disorders) | 5
Allergic reaction (Immune system disorders) | 2
Immune system disorders - Other, specify: Facial Flushing (Immune system disorders) | 1
Immune system disorders - Other, specify: lower back pain/raised rash (Immune system disorders) | 1
Bronchial infection (Infections and infestations) | 1
Infections and infestations - Other, specify: Bronchitis (Infections and infestations) | 1
Infections and infestations - Other, specify: Infection with Grade 3 (Infections and infestations) | 1
Infections and infestations - Other, specify: Upper Respiratory Infec (Infections and infestations) | 1
Infections and infestations - Other, specify: oral (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Arterial injury (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 5
Creatinine increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 1
Weight gain (Investigations) | 3
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 16
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: rig (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 28
Headache (Nervous system disorders) | 9
Nervous system disorders - Other, specify: Paresthesia (Nervous system disorders) | 1
Oculomotor nerve disorder (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 8
Trigeminal nerve disorder (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 5
Bladder spasm (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: Dysuria (Renal and urinary disorders) | 5
Renal and urinary disorders - Other, specify: Hematuria (Renal and urinary disorders) | 3
Urinary frequency (Renal and urinary disorders) | 6
Urinary incontinence (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: Pha (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: Upp (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: bro (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 5
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 27
Dry skin (Skin and subcutaneous tissue disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Nail loss (Skin and subcutaneous tissue disorders) | 5
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Skin and subcutaneous tissue disorders - Other, specify: Dermatology, (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: Inflamation (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: Vitiligo (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: rash (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: thinning ski (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 2
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 7
Thromboembolic event (Vascular disorders) | 1
Vascular disorders - Other, specify: Bleeding, rectal with bowel move (Vascular disorders) | 1
Vascular disorders - Other, specify: bronchitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes